CLINICAL TRIAL: NCT04254783
Title: A Phase 1 Study to Evaluate the Effect of Multiple IV Infusions of Risankizumab on the Pharmacokinetics of Cytochrome P450 Substrates Administered Orally in Subjects With Moderately to Severely Active Ulcerative Colitis or Crohn's Disease
Brief Title: A Study to Evaluate the Effect of Intravenous (IV) Infusions of Risankizumab on Pharmacokinetics of Cytochome P450 Substrates in Adult Participants With Moderately to Severely Active Ulcerative Colitis or Crohn's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M19-974; 2019-003684-22 (EudraCT Number)
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Ulcerative Colitis (UC); Crohn's Disease
Keywords: Ulcerative Colitis (UC); Crohn's Disease; Risankizumab; SKYRIZI; ABBV-066; Cytochrome P450
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — risankizumab; Cytochrome P-450 Enzyme System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cytochrome P450 (CYP) + Risankizumab (Experimental): In Period 1, participants will receive single oral dose of Cytochrome P450 (CYP) substrates on Day 1. In Period 2, three IV doses of risankizumab on Days 1, 29 and 57, followed by single oral dose of CYP substrates on Day 64 will be administered.
  Interventions: Drug: Risankizumab; Drug: Cytochrome P450 (CYP) Substrates

INTERVENTIONS:
Drug: Risankizumab — Intravenous (IV) infusion
  Other Names: SKYRIZI; ABBV-066
Drug: Cytochrome P450 (CYP) Substrates — Tablet: Oral; CYP Substrates: midazolam, caffeine, warfarin, vitamin K, omeprazole and metoprolol

SUMMARY:
Ulcerative colitis (UC) is a type of inflammatory bowel disease that causes inflammation and bleeding from the lining of the rectum and colon (large intestine).Crohn's disease (CD) is a long-lasting condition causing inflammation that can affect any part of the gut. CD may cause tiredness, loose stools with or without bleeding, abdominal pain, weight loss, and fever. This study will evaluate the effect of repeated infusions of risankizumab on the pharmacokinetics of sensitive probe substrates of Cytochrome P450 (CYP) enzymes in participants with moderately to severely active UC or CD.

Risankizumab is an investigational drug being developed to treat trial participants with inflammatory diseases such as UC and CD. The study is split into two periods. In Period 1, participants will receive single oral doses of CYP sensitive probes and in Period 2, participants will receive risankizumab followed by single oral doses of CYP sensitive probes. Around 20 adult participants with moderately to severely active CD or UC will be enrolled in the study across multiple sites worldwide.

In Period 1, participants will receive oral doses of CYP sensitive probes on Day 1. In Period 2, participants will receive risankizumab by intravenous (IV) infusion on Days 1, 29 and 57 followed by oral CYP sensitive probes on Day 64.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests and checking for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of UC or CD for at least 3 months prior to Day -1 (baseline). Appropriate documentation of biopsy results consistent with the diagnosis of CD or UC, in the assessment of the gastroenterologist, must be available.
* Moderately to severely active CD or UC.
* Must have demonstrated intolerance or inadequate response to one or more of the following categories of drugs: aminosalicylates, oral locally acting steroids, systemic steroids, immunomodulators, and/or approved biologic therapies.
* Participant must agree to not use any known inhibitors or inducers of cytochrome P450 within 1 month or 5 half-lives, whichever is greater before each administration of the cocktail probe and until the last pharmacokinetic sample is collected, 7 days after the intake of each probe cocktail.

Exclusion Criteria:

* History of any clinically significant sensitivity or allergy to any medication or food.
* History of or active medical condition(s) or surgical procedure(s) that might affect gastrointestinal motility, pH, or absorption (e.g., celiac disease, gastroparesis, cholecystectomy, vagotomy).
* Positive for COVID-19 infection signs and symptoms.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Midazolam | Up to 71 Days
  Maximum observed plasma concentration (Cmax) of Midazolam
Time to Maximum Observed Plasma Concentration (Tmax) of Midazolam | Up to 71 Days
  Time to maximum plasma concentration (Tmax) of Midazolam
Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to Time of the Last Measurable Concentration (AUCt) of Midazolam | Up to 71 Days
  Area Under the Plasma Concentration-time Curve (AUC) from time 0 to time of the last measurable concentration
AUC From Time 0 to Infinity (AUCinf) of Midazolam | Up to 71 Days
  Area Under the Plasma Concentration-time Curve (AUC) from time 0 to infinity
Terminal Phase Elimination Rate Constant (β) of Midazolam | Up to 71 Days
  Terminal phase elimination rate constant (β) for Midazolam
Terminal Phase Elimination Half-Life (t1/2) of Midazolam | Up to 71 Days
  Terminal phase elimination half-life (t1/2) of Midazolam
Maximum Observed Plasma Concentration (Cmax) of Caffeine | Up to 71 Days
  Maximum observed plasma concentration (Cmax) of Caffeine
Time to Maximum Observed Plasma Concentration (Tmax) of Caffeine | Up to 71 Days
  Time to maximum plasma concentration (Tmax) of Caffeine
Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to Time of the Last Measurable Concentration (AUCt) of Caffeine | Up to 71 Days
  Area Under the Plasma Concentration-time Curve (AUC) from time 0 to time of the last measurable concentration
AUC From Time 0 to Infinity (AUCinf) of Caffeine | Up to 71 Days
  Area Under the Plasma Concentration-time Curve (AUC) from time 0 to infinity
Terminal Phase Elimination Rate Constant (β) of Caffeine | Up to 71 Days
  Terminal phase elimination rate constant (β) for Caffeine
Terminal Phase Elimination Half-Life (t1/2) of Caffeine | Up to 71 Days
  Terminal phase elimination half-life (t1/2) of Caffeine
Maximum Observed Plasma Concentration (Cmax) of Warfarin | Up to 71 Days
  Maximum observed plasma concentration (Cmax) of Warfarin
Time to Maximum Observed Plasma Concentration (Tmax) of Warfarin | Up to 71 Days
  Time to maximum plasma concentration (Tmax) of Warfarin
Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to Time of the Last Measurable Concentration (AUCt) of Warfarin | Up to 71 Days
  Area Under the Plasma Concentration-time Curve (AUC) from time 0 to time of the last measurable concentration
AUC From Time 0 to Infinity (AUCinf) of Warfarin | Up to 71 Days
  Area Under the Plasma Concentration-time Curve (AUC) from time 0 to infinity
Terminal Phase Elimination Rate Constant (β) of Warfarin | Up to 71 Days
  Terminal phase elimination rate constant (β) for Warfarin
Terminal Phase Elimination Half-Life (t1/2) of Warfarin | Up to 71 Days
  Terminal phase elimination half-life (t1/2) of Warfarin
Maximum Observed Plasma Concentration (Cmax) of Omeprazole | Up to 71 Days
  Maximum observed plasma concentration (Cmax) of Omeprazole
Time to Maximum Observed Plasma Concentration (Tmax) of Omeprazole | Up to 71 Days
  Time to maximum plasma concentration (Tmax) of Omeprazole
Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to Time of the Last Measurable Concentration (AUCt) of Omeprazole | Up to 71 Days
  Area Under the Plasma Concentration-time Curve (AUC) from time 0 to time of the last measurable concentration
AUC From Time 0 to Infinity (AUCinf) of Omeprazole | Up to 71 Days
  Area Under the Plasma Concentration-time Curve (AUC) from time 0 to infinity
Terminal Phase Elimination Rate Constant (β) of Omeprazole | Up to 71 Days
  Terminal phase elimination rate constant (β) for Omeprazole
Terminal Phase Elimination Half-Life (t1/2) of Omeprazole | Up to 71 Days
  Terminal phase elimination half-life (t1/2) of Omeprazole
Maximum Observed Plasma Concentration (Cmax) of Metoprolol | Up to 71 Days
  Maximum observed plasma concentration (Cmax) of Metoprolol
Time to Maximum Observed Plasma Concentration (Tmax) of Metoprolol | Up to 71 Days
  Time to maximum plasma concentration (Tmax) of Metoprolol
Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to Time of the Last Measurable Concentration (AUCt) of Metoprolol | Up to 71 Days
  Area Under the Plasma Concentration-time Curve (AUC) from time 0 to time of the last measurable concentration
AUC From Time 0 to Infinity (AUCinf) of Metoprolol | Up to 71 Days
  Area Under the Plasma Concentration-time Curve (AUC) from time 0 to infinity
Terminal Phase Elimination Rate Constant (β) of Metoprolol | Up to 71 Days
  Terminal phase elimination rate constant (β) for Metoprolol
Terminal Phase Elimination Half-Life (t1/2) of Metoprolol | Up to 71 Days
  Terminal phase elimination half-life (t1/2) of Metoprolol

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (6):
- United States (4):
  - Southern California Res. Ctr. /ID# 216257, Coronado, California
  - University Clinical Research /ID# 216823, DeLand, Florida
  - Atlantic Medical Research Group /ID# 227465, Margate, Florida
  - Clinical Trials of Texas, Inc /ID# 216277, San Antonio, Texas
- Charite Research Organisation GmbH /ID# 218646, Berlin, Germany
- The Chaim Sheba Medical Center /ID# 223959, Ramat Gan, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D'Cunha R, Azam T, Kalabic J, Anschutz T, Lahat A, Pang Y. Evaluation of the Effect of Risankizumab on the Pharmacokinetics of Cytochrome P450 Substrates in Patients with Moderately to Severely Active Ulcerative Colitis or Crohn's Disease. Clin Pharmacokinet. 2025 Jan;64(1):143-154. doi: 10.1007/s40262-024-01462-4. Epub 2024 Dec 21. PMID 39707077
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=M19-974#additional-resources-section